CLINICAL TRIAL: NCT04164147
Title: Comparison of the Persona Medial Congruent Retained Posterior-Cruciate Ligament vs. Persona Posterior-stabilized vs. NexGen Posterior-Stabilized Total Knee Arthroplasty a Randomised Controlled Trial
Brief Title: Persona MC Retained PCL vs. Persona Posterior-stabilized vs. NexGen PS
Acronym: Persona TKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Head of the Department of Orthopedic and Rehabilitation, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WarszawMU
Record Dates: First submitted 2019-10-31; First posted 2019-11-15 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis; Knee Arthritis; Joint; Arthrosis, Primary
Keywords: Total Knee Arthroplasty; Nexgen; Persona; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee; Tomography, X-Ray Computed; Biomechanical Phenomena

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will not be informed which type of prosthesis was used in their particular case.
  Outcomes Assessor will not be informed which type of prosthesis was used in particular patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NexGen (Active Comparator): Patients undergoing total knee replacement for treatment of primary knee ostearthritis with use of Zimmer Biomet NexGen prosthesis
  Interventions: Procedure: Total knee replacement; Diagnostic Test: CT scan; Diagnostic Test: Biomechanics; Device: one of the Persona MC Retained PCL, Persona MC Sacrificed PCL and NexGen PS total knee implant
- Persona MC Retained PCL (Active Comparator): Patients undergoing total knee replacement for treatment of primary knee ostearthritis with use of Zimmer Biomet Persona MC Retained PCL prosthesis
  Interventions: Procedure: Total knee replacement; Diagnostic Test: CT scan; Diagnostic Test: Biomechanics; Device: one of the Persona MC Retained PCL, Persona MC Sacrificed PCL and NexGen PS total knee implant
- Persona MC Sacrificed PCL (Active Comparator): Patients undergoing total knee replacement for treatment of primary knee ostearthritis with use of Zimmer Biomet Persona MC Sacrificed PCL prosthesis
  Interventions: Procedure: Total knee replacement; Diagnostic Test: CT scan; Diagnostic Test: Biomechanics; Device: one of the Persona MC Retained PCL, Persona MC Sacrificed PCL and NexGen PS total knee implant

INTERVENTIONS:
Procedure: Total knee replacement — Participant will undergo total knee replacement performed via anterior parapatellar approach with either Posterior Cruciate Ligament sacrificing or retaining implant
Diagnostic Test: CT scan — CT scans of the affected knee joint before and after the surgical procedure
Diagnostic Test: Biomechanics — Participants will be asked to perform biomechanical assesment before and following surgery at baseline, 6-8 weeks and 6-months postoperatively
Device: one of the Persona MC Retained PCL, Persona MC Sacrificed PCL and NexGen PS total knee implant — Participant are randomly allocated to receive one of the Persona MC Retained PCL, Persona MC Sacrificed PCL and the NexGen PS total knee implant for treatment of end-stage knee osteoarthritis.

SUMMARY:
This study compares and evaluates differences in movement analysis, patient-reported outcome and radiological assesment between patients undergoing total knee arthroplasty with use of either Zimmer Biomet NexGen and Zimmer Biomet PERSONA

DETAILED DESCRIPTION:
Osteoarthritis causes the joints to become painful and stiff. Osteoarthritis of the knee is a common condition that is expected to be a lot more frequent in the next two decades. As a consequence, an increase of total knee replacement surgery is predicted. Total knee replacement surgery is offered when knee pain and stiffness caused by osteoarthritis can no longer be managed and these symptoms significantly impact on an individual's normal activities of daily living. Most total knee replacements are successful but up to 34% of all patients have poor functional outcomes following surgery. This leaves affected people at a greater risk of reduced physical activity and thus impacts longer-term general health. Poor outcomes are therefore of importance to patients and have a considerable financial and service-provision impact on National Health Service (NHS) care. While patient-related characteristics and their relationship to patient outcomes have been identified, few studies have been undertaken to determine how kinematic outcomes (how the prosthetic knee moves) are related to functional outcome and patient satisfaction. The kinematic outcome of a total knee replacement is hypothesised to relate to both the structural design (shape) of the implant and the surgical procedure itself. To date, no studies have investigated the kinematic outcomes of different total knee replacement prosthesis designs through a range of typical activities of everyday mobility (functional outcomes). Whilst it is known that long term success of total knee replacement depends largely upon correct alignment of the prosthesis components during surgery, no studies have looked at the anatomical alignments of the osteoarthritic knee prior to undergoing surgery (using Computerised Tomography (CT) scanning). The aim of the study is to examine relationships between movement analysis (kinematic and functional outcomes), patient reported outcome measures (PROMS) and CT measurement, both pre- and post-operatively, between two knee prosthesis including one that has been designed to improve functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Listed for a primary total knee replacement (TKR) at the Orthopaedic and Rehabilitation Department Medical University of Warsaw
2. Indication for the TKR is primary osteoarthritis of the knee joint involving one or more compartments
3. Aged 18 or over
4. Patient willing to provide full informed consent to the trial

Exclusion Criteria:

1. Listed for a single-stage bilateral TKR procedure
2. Severe symptoms in the contralateral knee so as to require staged bilateral knee replacements within 6 months of the primary procedure
3. Fixed flexion deformity of 15 degrees or greater who will require excessive resection of the distal femur
4. Clinically assessed uncorrectable varus/valgus deformity of 15 degrees or greater
5. Any co-morbidity which, in the opinion of the investigator, is severe enough to present an unacceptable risk to the patient's safety
6. Inflammatory arthritis
7. Previous septic arthritis in the affected knee joint
8. Previous surgery to the collateral ligaments of the affected knee
9. A contralateral total knee replacement that has been implanted less than one year from the date of consultation
10. A contralateral total knee replacement that is severely painful
11. Patients on warfarin or novel oral anticoagulants (NOACs)
12. Will not be resident in the catchment area for at least 6 months post-surgery
13. Undertaking the surgery as a private patient
14. Patients who, in the opinion of the clinical staff, do not have capacity to consent
15. Patients who are pregnant
16. Unable to understand written and spoken Polish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in patients reported outcome measures - Oxford Knee Score (OKS) | baseline (preoperatively) and 6-months postoperatively
  To explore differences between outcome in patients treated with use of with Nexgen and Persona prosthesis. Results range from 0 to 48, with higher scores corresponding to better outcomes.

SECONDARY OUTCOMES:
Changes in patients reported outcome measures - Oxford Knee Score (OKS) | 1 week and 6-8 weeks post-operatively
  To explore differences between outcome in patients treated with use of with Nexgen and Persona prosthesis. Results range from 0 to 48, with higher scores corresponding to better outcomes.
Changes in patients reported outcomes - Oxford Knee Score Activity & Participation Questionnaire (OKS_APQ) | 1 week, 6-8 weeks and 6 months post- operatively
  To explore differences in higher levels of activity and social participation
Changes in patients reported outcomes - EuroQol (EQ- 5D-5L) | 1 week, 6-8 weeks and 6 months post- operatively
  To explore differences in quality of life
Changes in patients reported outcomes - Forgotten Joint Score (FJS) | 6-8 weeks and 6 months post-operatively
  To explore differences in patient's ability to forget about a joint as a result of successful treatment. Results range from 0 to 100, with higher scores corresponding to better outcomes.
Changes in patients reported outcomes - UCLA (University of California) score | 6-8 weeks and 6 months post-operatively
  To explore differences in patient's physical activity. Results range from 0 to 10, with higher scores corresponding to better outcomes.
Changes in knee range of motion | preoperatively, 6-8 weeks and 6 months post-operatively
  To explore differences in range of motion (flexion and extension)
Changes in pain medication | 1 week, 6-8 weeks and 6 months post-operatively
  To asses evolution of post-operative knee pain
arthroplasty related complications | 1 week, 6-8 weeks and 6 months post-operatively
  To count and asses all complications that may occur during surgery and in postoperative period
arthroplasty revision surgeries | 1 week, 6-8 weeks and 6 months post-operatively
  To count and asses the reason of all revision surgeries that may occur during postoperative period
walking abilities | 6-8 weeks and 6 months post-operatively
  To asses "up and go" time
Length of hospital stay | from baseline to discharge from hospital ranging averagely from 1 up to 7 days postoperatively
  To measure number of days counting from surgery to the discharge
Biomechanical 3D miotion and emg walking outcomes | at baseline, 6-8 weeks and 6 months post-operatively
  Overground walking is measured using 3D Motion analysis and electromyography (EMG)
Radiological outcome on CT scans | at baseline preoperatively and 6-months postoperatively
  Rotational alignment of the total knee component is assessed by measuring the femoral antetorsion, Alignment of the total knee component is assessed by measuring the tibial tubercle-trochlear groove distance (TT-TG)
6- minute walking abilities | 6-8 weeks and 6 months post-operatively
  to asses pace and model of 6-minute walk
Biomechanical stair climbing outcomes | at baseline, 6-8 weeks and 6 months post-operatively
  Stair climbing and descending is measured using 3D Motion analysis and EMG
Biomechanical static balance outcomes | at baseline, 6-8 weeks and 6 months post-operatively
  Static balance is measured using a force plate
Biomechanical dynamic balance outcomes | at baseline, 6-8 weeks and 6 months post-operatively
  Dynamic balance is measured using a force plate and the modified Star Excursion Balance Test (mSEBT)
Leg muscle strength outcomes | at baseline, 6-8 weeks and 6 months post-operatively
  Leg muscle strength measured using maximal voluntary isometric contraction (MVIC) test of the hamstring and quadriceps muscles on both limbs.

CONTACTS AND LOCATIONS:
Overall Officials: Artur Stolarczyk, PhD, Study Director — Medical University of Warsaw
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maciag BM, Kordyaczny T, Jegierski D, Lapinski M, Dorocinska M, Zarnovsky K, Maciag GJ, Adamska O, Stolarczyk A. Differences in joint line level and posterior condylar offset during total knee replacement with use of gap-balancing and measured resection techniques-matched cohort study. BMC Musculoskelet Disord. 2023 Jul 25;24(1):610. doi: 10.1186/s12891-023-06722-1. PMID 37491199